CLINICAL TRIAL: NCT04810546
Title: Feasibility or Oral Lactoferrin to Prevent Iron Deficiency Anemia in Obese Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary Dawn Koenig, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-1297; R34HL155481 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-03-23 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Iron-deficiency; Pregnancy Anemia; Obesity
MeSH Terms: conditions — Anemia, Iron-Deficiency; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Jarrow Formulas Oral Bovine Lactoferrin Supplement (Experimental): Once daily Oral Lf (250mg). Women assigned to this group will be instructed to consume an oral Lf capsule one hour prior to their afternoon meal and two prenatal vitamin/mineral supplement gummies without iron with omega-3 fatty acids before bed from early second trimester (15 - 20 WG) up through delivery. Women are advised to consume the Lf prior to meals, given our team member Valenti's unpublished work shows its superior efficacy for improving iron and hematological parameters among pregnant women with hereditary thrombophilia versus when consumed with meals. The prenatal vitamin/mineral gummies will be a commercially available product (One-a-Day Women's Prenatal Gummies with omega-3 fatty acids, Bayer Healthcare, Whippany, NJ). Women in both groups will be advised to consume an iron-rich diet and provided a handout detailing foods rich in heme and non-heme iron.
  Interventions: Dietary Supplement: Jarrow Formulas Oral Bovine Lactoferrin Supplement
- Usual care (No Intervention): Women assigned to this group will be instructed to consume a commercially available prenatal vitamin/mineral supplement with iron and omega-3 fatty acids (Prenatal 1, Bayer Healthcare, Whippany, NJ) before bed from early second trimester (15-20 WG) through delivery. To minimize variability in prenatal vitamin/supplement use across the participants, we have opted to standardize the prenatal vitamin/mineral supplement by providing women in the usual care arm a supplement that is nutritionally like what is prescribed by the Center for Women's Health providers. Women will be advised to consume an iron-rich diet and provided a handout describing foods rich in heme and non-heme iron.

INTERVENTIONS:
Dietary Supplement: Jarrow Formulas Oral Bovine Lactoferrin Supplement — Lactoferrin (Apolactoferrin) 250mg contains ~17.6 mg/100g of iron
  Arms: Jarrow Formulas Oral Bovine Lactoferrin Supplement

SUMMARY:
Maternal iron deficiency anemia is associated with maternal and infant mortality, spontaneous preterm birth, maternal postpartum hemorrhage, and neurocognitive defects in the neonate. Therefore, preventing maternal iron deficiency anemia in at-risk women is critical. Obese pregnant women have greater systemic inflammation and circulating hepcidin levels compared to nonobese pregnant women. This phenotype implies obese pregnant women have decreased iron bioavailability and may be less responsive to oral iron supplementation because hepcidin is a negative regulator of dietary iron absorption, suggesting alternative interventions are needed to optimize their iron status in pregnancy. There is increasing evidence that consuming the oral bovine lactoferrin (bLf) can enhance dietary iron absorption by promoting an anti-inflammatory immune response and hepcidin suppression, indicating this intervention may be beneficial to pregnant obese women at risk for iron deficiency anemia. The primary goal of this study is to test the feasibility and acceptability of this low-cost, safe, innovative approach to optimizing maternal iron status in obese women at risk of iron deficiency anemia (Hb 11.0 - 12.0 g/dL (first trimester)/10.5 - 11.5 g/dL (second trimester) for non-Black women and 10.2 - 11.2 g/dL (first trimester)/9.7 -- 10.7 g/dL (second trimester) for Black women) from 15-20 weeks of gestation (WG) until the time of labor. The investigators will explore effects on maternal and neonatal iron status and Hb and changes to maternal systemic inflammation and circulating hepcidin. This study is an essential first step toward evaluating if daily oral bLf is an efficacious, safe, inexpensive, and scalable clinical strategy for the prevention of maternal iron deficiency anemia and its related complications in at-risk women.

ELIGIBILITY:
Inclusion Criteria:

* naturally conceived, single pregnancy
* at risk of IDA [Hb 11.0 - 12.0 g/dL (first trimester)/10.5 - 11.5 g/dL (second trimester) for non-Black women and 10.2 - 11.2 g/dL (first trimester)/9.7 -- 10.7 g/dL (second trimester) for Black women]42 based on new OB complete blood count (CBC) results obtained from the EMR
* 18 - 45 years old
* pre-conception BMI ≥ 30.0 kg/m2 [based on measured height in EMR and recent pre-conception weight (within 3 months of pregnancy) from EMR if available or self-reported]; < 20 WG
* fluency in English to provide consent and complete study procedures;
* ability to provide consent
* ownership of a smartphone (currently more than 90% of our patient population at the Center for Women's Health)

Exclusion Criteria:

* birth, or other pregnancy in the previous 12 months
* IDA requiring high dose supplemental iron
* allergy to milk proteins or wheat
* vegan (due to content of the supplements)
* recent blood transfusion
* previously diagnosed type 1 or type 2 diabetes
* autoimmune disorder (e.g., rheumatoid arthritis)
* inflammatory bowel disease
* premature rupture of membranes or chorioamnionitis
* previous spontaneous preterm birth
* current bacterial or viral infection
* history of bariatric surgery
* malabsorptive disease
* current hyperemesis
* current eating disorder
* hematologic disorder or trait carrier (e.g., hemochromatosis, β-thalassemia)
* current tobacco, alcohol or illicit drug use (including marijuana)
* regular use of medications that may interfere with nutrient absorption
* unstable housing, first trimester PHQ-9 score > 10, and/or a recent traumatic event (e.g., death of a significant other or parent) may make it difficult to comply with the interventions, hence these women will also be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Understand feasibility via recruitment and retention rates | Recruitment duration- approximately 3 years
  We will collect detailed records of the number of women eligible and then referred by Center for Women's Health clinical staff to the research team. We will also track the number of referred women approached (by phone & in person) by our research team for enrollment and the number of women who decline and their reasons for non-enrollment. Once a woman is enrolled in the study, attendance at study visits, completeness of data, and overall and treatment specific loss to follow-up/withdrawal will be closely monitored. Women who voluntarily withdraw will be asked to provide reasons for revoking their enrollment. Rates of enrollment and retainment are key feasibility outcomes. To facilitate recruitment and retention, transportation and participation monetary incentives will be provided. Data will be evaluated to determine feasibility of this kind of reasearch
Measure participant adherence | 8 months
  For both study arms, the Pillsy smart bottle, phone app, and researcher interface configured, tested and finalized in Aim 1 will be used to optimize adherence. The smart bottle will send reminders (i.e., the pill bottle rings and lights up) at a time selected by the participant congruent with their intervention arm assignment (e.g., at bedtime). Use of the Pillsy app will allow for "real-time" tracking of the participant's adherence through the HIPAA-compliant researcher interface. If a participant is non-adherent for two consecutive days additional alerts (e.g., text messages) will be triggered through the research interface two-way communication feature, and study staff will make contact (i.e., telephone/text/email). Hand pill counts will also be performed by UIC Investigational Drug Service. Smart bottles will generate individual reports detailing how many pills were taken and when. A report detailing dates and times of pills being taken will be used to measure adherence
Determine preliminary efficacy on maternal inflammation | baseline
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at baseline with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%. Expected results: We expect significantly lower IL-6 at 19-24 weeks gestation that is maintained through delivery in women randomized to oral Lf compared with control.
Determine preliminary efficacy on maternal inflammation | month 3
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at 23-28 weeks gestation (month 3) with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%. Expected results: We expect significantly lower IL-6 at 19-24 weeks gestation that is maintained through delivery in women randomized to oral Lf compared with control.
Determine preliminary efficacy on maternal inflammation | month 5
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at 31-36 weeks gestation (month 5) with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%. Expected results: We expect significantly lower IL-6 at 19-24 weeks gestation that is maintained through delivery in women randomized to oral Lf compared with control.
Determine preliminary efficacy on maternal inflammation | labor (~month 8)
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at admittance for labor and delivery with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%. Expected results: We expect significantly lower IL-6 at 19-24 weeks gestation that is maintained through delivery in women randomized to oral Lf compared with control.
Determine preliminary efficacy on maternal iron and hematological markers. | baseline
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at baseline
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | baseline
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at baseline
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | baseline
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at baseline
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | baseline
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at baseline
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 1 month
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 1 month
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 1 month
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 1 month
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 2 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 2 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 2 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 2 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 3 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 3 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 3 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 3 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at monthly.
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 4 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 4 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 4 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 4 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 5 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 5 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 5 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 5 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 6 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 6 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 6 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 6 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | 7 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | 7 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | 7 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | 7 months
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood monthly
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal iron and hematological markers. | delivery (~8 months)
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at admittance for delivery.
  • Ferritin & Iron. Maternal ferritin and iron will be measured in serum by immunoassay and spectrophotometry by a local commercial lab
Determine preliminary efficacy on maternal iron and hematological markers. | delivery (~8 months)
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at admittance for delivery.
  • sTFR. Maternal sTFR will be measured in serum using a commercially available immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on maternal iron and hematological markers. | delivery (~8 months)
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at admittance for delivery.
  • Calculated Total Body Iron (TBI). Maternal TBI will be calculated from sTFR and serum ferritin using an equation developed by Cook and colleagues.
Determine preliminary efficacy on maternal iron and hematological markers. | delivery (~8 months)
  Maternal iron status and hematological parameters will be assessed from antecubital non-fasting blood at admittance for delivery.
  • Complete Blood Count (CBC). Maternal CBC with differential will be measured in whole blood by electronic cell sizing/counting/cytometry/microscopy by a local commercial lab). Hb is the primary clinical outcome for the trial given it is the most commonly assessed iron/hematological status marker in pregnancy.
Determine preliminary efficacy on maternal hematological markers. | Baseline
  Maternal Hepcidin. Maternal hepcidin will be measured in serum at baseline with a commercially available ELISA. The minimum level of detection for the assay is 2.5 ng/mL.
Determine preliminary efficacy on maternal hematological markers. | Baseline
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at baseline with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%.
Determine preliminary efficacy on maternal hematological markers. | Baseline
  . Maternal Erythropoietin. Erythropoiesis is a negative regulator of hepcidin. Maternal erythropoietin will be measured in serum at baseline with a commercially available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 2.6%.
Determine preliminary efficacy on maternal hematological markers. | 3 months
  Maternal Hepcidin. Maternal hepcidin will be measured in serum at 3 months with a commercially available ELISA. The minimum level of detection for the assay is 2.5 ng/mL.
Determine preliminary efficacy on maternal hematological markers. | 3 months
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at 3 months with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%.
Determine preliminary efficacy on maternal hematological markers. | 3 months
  Maternal Erythropoietin. Erythropoiesis is a negative regulator of hepcidin. Maternal erythropoietin will be measured in serum at 3 months with a commercially available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 2.6%.
Determine preliminary efficacy on maternal hematological markers. | 5 months
  Maternal Hepcidin. Maternal hepcidin will be measured in serum at 5 months with a commercially available ELISA. The minimum level of detection for the assay is 2.5 ng/mL.
Determine preliminary efficacy on maternal hematological markers. | 5 months
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at 5 months with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%.
Determine preliminary efficacy on maternal hematological markers. | 5 months
  Maternal Erythropoietin. Erythropoiesis is a negative regulator of hepcidin. Maternal erythropoietin will be measured in serum at 5 months with a commercially available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 2.6%.
Determine preliminary efficacy on maternal hematological markers. | Delivery (~8 months)
  Maternal Hepcidin. Maternal hepcidin will be measured in serum at admittance for labor and delivery with a commercially available ELISA. The minimum level of detection for the assay is 2.5 ng/mL.
Determine preliminary efficacy on maternal hematological markers. | Delivery (~8 months)
  Maternal IL-6. Inflammation, specifically the pro-inflammatory cytokine IL-6, is a positive regulator of hepcidin. Maternal IL-6 will be measured in serum at admittance for labor and delivery with a commercially-available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 5.7%.
Determine preliminary efficacy on maternal hematological markers. | Delivery (~8 months)
  Maternal Erythropoietin. Erythropoiesis is a negative regulator of hepcidin. Maternal erythropoietin will be measured in serum at admittance for labor and delivery with a commercially available ELISA (R&D Systems, Minneapolis, MN). Our lab's intra-assay CV is 2.6%.
Determine preliminary efficacy on neonatal iron and hematological markers. | Delivery (~8 months)
  Neonatal cord iron status and hematologic parameters will be assessed from venous umbilical cord blood obtained bedside following delivery of the placenta. Even with delayed umbilical cord-clamping, we can successfully obtain 40-50 milliliters of umbilical venous cord blood.
  • Cord Ferritin & Iron. Cord ferritin and iron will be measured in serum by immunoassay and spectrophotometry at a local commercial lab (Quest Diagnostics, Wood Dale, IL).
Determine preliminary efficacy on neonatal iron and hematological markers. | Delivery (~8 months)
  Neonatal cord iron status and hematologic parameters will be assessed from venous umbilical cord blood obtained bedside following delivery of the placenta. Even with delayed umbilical cord-clamping, we can successfully obtain 40-50 milliliters of umbilical venous cord blood.
  • Cord sTFR. Cord sTFR will be measured with an immunoassay (ELISA) (R&D Systems, Minneapolis, MN). Our lab's intra-assay coefficient of variation (CV) for this kit is 5.3%.
Determine preliminary efficacy on neonatal iron and hematological markers. | Delivery (~8 months)
  Neonatal cord iron status and hematologic parameters will be assessed from venous umbilical cord blood obtained bedside following delivery of the placenta. Even with delayed umbilical cord-clamping, we can successfully obtain 40-50 milliliters of umbilical venous cord blood.
  • Cord TBI. Cord TBI will be calculated from cord sTFR and serum ferritin using a published equation.
Determine preliminary efficacy on neonatal iron and hematological markers. | Delivery (~8 months)
  Neonatal cord iron status and hematologic parameters will be assessed from venous umbilical cord blood obtained bedside following delivery of the placenta. Even with delayed umbilical cord-clamping, we can successfully obtain 40-50 milliliters of umbilical venous cord blood.
  • Cord CBC. Cord CBC with differential, which includes Hb, will be measured by electronic cell sizing/counting/cytometry/microscopy at a local commercial lab (Quest Diagnostics, Wood Dale, IL).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dawn Koenig, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States